CLINICAL TRIAL: NCT05913310
Title: A Randomized Controlled Study of Kui-Yuan Chewable Tablets in the Treatment of Hyperuricemia
Brief Title: Efficacy and Safety of Kui-Yuan Chewable Tablets in Patients With Hyperuricemia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Quan Jiang (Other)
Responsible Party: Sponsor-Investigator, Quan Jiang, chief physician, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Organization: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023023P7A01
Record Dates: First submitted 2023-06-09; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Hyperuricemia
Keywords: Hyperuricemia; Kui-Yuan Chewable; Randomized controlled trial
MeSH Terms: conditions — Hyperuricemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kui-Yuan Chewable Tablets (Active Comparator)
  Interventions: Drug: Kui-Yuan Chewable Tablets
- Placebo of Kui-Yuan Chewable Tablets (Placebo Comparator)
  Interventions: Drug: Placedo of Kui-Yuan Chewable Tablets

INTERVENTIONS:
Drug: Kui-Yuan Chewable Tablets — Kui-Yuan chewable tablets are the optimal ingredients found in sunflower dish that can reduce uric acid and anti-gout, including flavonoids, Coumarin (including scopolamine) and phenolic acids.
  Arms: Kui-Yuan Chewable Tablets
Drug: Placedo of Kui-Yuan Chewable Tablets — Placedo of Kui-Yuan Chewable Tablets are composed of L-arabinose, food starch and a few auxiliary materials.
  Arms: Placebo of Kui-Yuan Chewable Tablets

SUMMARY:
This study is a multi-center, randomized, double-blinded, controlled trial with two parallel arms. The aim of the study is to evaluate efficacy and safety of Kui-Yuan chewable tablets in patients with hyperuricemia.

ELIGIBILITY:
Inclusion Criteria:

* Blood uric acid level>7.0mg/dL (420 μmol/L)
* The participants did not experience any acute gout attacks before treatment
* The ECG of the participants was normal before treatment

Exclusion Criteria:

* Secondary Hyperuricemia caused by kidney disease, blood disease, or taking certain drugs, tumor radiotherapy and chemotherapy, organ transplantation, etc
* Those who have used allopurinol, probenecid, benzbromarone, febuxostat or traditional Chinese medicine with uric acid lowering effect within 4 weeks before enrollment
* Those who had a history of cardiovascular and cerebrovascular diseases such as stroke, TIA, MI, HF (NYHA grade II-IV), and coronary artery surgery (such as angioplasty, stent implantation, bypass grafting, etc.)
* Those who had a history of gastrointestinal ulcers or gastrointestinal bleeding
* Active liver disease or abnormal liver function, ALT and AST are more than 3 times the upper limit of normal
* Glomerular filtration rate (eGFR)<30mL/min/1.73m2
* Those who are allergic or intolerant to any component in Kui-Yuan chewable tablets and placebo
* Those who had other autoimmune diseases
* Those who are taking or need to take aspirin, other salicylic acids, heparin, Dicoumarol and other anticoagulants and antiplatelet aggregation drugs
* Those who taking Diuretic
* Those who had a history of alcohol or drug dependence, or those who require long-term daily use of painkillers for any reason
* Pregnancy, lactation, or planned pregnancy within 3 months after the last study medication

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Proportion of sUA levels below 420 μmol/L | 3 months
  Proportion of participants maintaining sUA levels below 420 μmol/L at the third month

SECONDARY OUTCOMES:
Proportion of sUA levels below 360 μmol/L | 3 months
  Proportion of participants maintaining sUA levels below 360 μmol/L at the third month
The number of gout attacks | 3 months
  The number of gout attacks from baseline to month 3
Proportion of gout attacks | 3 months
  Proportion of participants reporting gout attacks from baseline to month 3
Percentage change in sUA levels | 3 months
  Percentage change of participants in sUA levels from baseline to each visit
Changes in BMI | 3 months
  Changes in participants' BMI from baseline to the third month (combined with obesity)
Changes in blood pressure levels | 3 months
  Changes in participants' blood pressure levels from baseline to the third month (combined with hypertension)
Changes in blood lipid levels | 3 months
  Changes in participants' blood lipid levels from baseline to the third month (combined with hyperlipidemia)
Changes in fasting blood glucose levels | 3 months
  Changes in participants' fasting blood glucose levels from baseline to the third month (combined with diabetes)

IPD SHARING:
Plan to Share IPD: No